CLINICAL TRIAL: NCT05260970
Title: The Effect of Rectus Muscle Re-approximation on Postoperative Pain Among Primigravida Singleton Pregnancies Who Underwent Elective Cesarean Section: A Randomized Prospective Trial
Brief Title: The Effect of Rectus Muscle Re-approximation at Cesarean Delivery on Postoperative Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Orkun Cetin, Associate Professor, Balikesir University
Other Study IDs: rectus1
Record Dates: First submitted 2022-01-24; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Suturing of Rectus Muscle at Cesarean Section
Keywords: Cesarean section; Rectus Muscle; Rectus Muscle Re-approximation; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- undergoing rectus muscle reapproximation: Primigravida Singleton Pregnancies Who Underwent Elective Cesarean Section with rectus muscle reapproximation procedure
  Interventions: Procedure: Rectus muscle reapproximation at cesarean section
- not undergoing rectus muscle reapproximation: Primigravida Singleton Pregnancies Who Underwent Elective Cesarean Section without rectus muscle reapproximation procedure

INTERVENTIONS:
Procedure: Rectus muscle reapproximation at cesarean section — Rectus muscle reapproximation: Continuous Suturing of rectus muscles with 2.0 Vicryl (Ethicon) at Cesarean section.
  Groups: undergoing rectus muscle reapproximation

SUMMARY:
The Effect of Rectus Muscle Re-approximation on Postoperative Pain Among Primigravida Singleton Pregnancies Who Underwent Elective Cesarean Section: A Randomized Prospective Trial.

Cesarean section is the most common surgical procedure performed in women in all around the world. Cesarean delivery rate has increased dramatically worldwide but there is still debate about the optimum operative technique of cesarean section.

Rectus muscle reapproximation, or suturing of the rectus muscles, is performed by many obstetricians in several countries, presumably to reduce the risk of persistent rectus muscle diastasis. However, there was a few studies about the short and long term effects of rectus muscle reapproximation in the literature.

On this account, the investigators aimed to design a randomized prospective trial about the effect of rectus muscle re-approximation on postoperative pain among primigravida singleton pregnancies who underwent elective cesarean section.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial conducted at Balikesir University Medical Faculty Department of Obstetrics and Gynecology at Balikesir, Turkey between January 2021 and March 2022. The singleton pregnant women undergoing scheduled primary cesarean section who are not in labor and consented to the trial are randomly assigned to receive rectus muscle reapproximation versus no reapproximation.

Gestational age is detected by the first day of last menstrual period and confirmed by first trimester ultrasonography measurements. The pregnant women who recruited this study would have no maternal accompanying conditions, such as hypertensive disorders of pregnancy, preterm rupture of membranes, Type 1 diabetes mellitus, gestational diabetes mellitus, reno-vascular disorders, sickle-cell anemia, collagen-vascular diseases, hereditary or acquired thrombophilia, congenital abnormalities and multiple gestations. Randomization would be conducted through sequentially numbered opaque envelopes generate by a study nurse in blocks through a random numbers table, in a 1:1 ratio.

Surgical techniques at cesarean section are standardized within the study and included closure of the parietal peritoneum and one-layer uterine closure. For women randomized to rectus muscle reapproximation, surgeons will use 2.0 Vicryl (Ethicon) for continuous suturing to reapproximate the rectus muscles. All surgeries were performed by an attending physician and a resident physician.Intraoperative analgesia was standardized to spinal anesthesia. Postoperative pain management is standardized by using our clinic's postoperative cesarean section protocol.Patients with pain unresponsive to the aforementioned treatment could receive opioids as necessary. Visual analog scale (VAS)scores are assessed through inperson interview in the hospital by a member of the study team at 24 and 48 hours after cesarean section.Total opioid use, total milligrams of nonsteroid antiinflammatory drugs (NSAIDs) and acetaminophen use are also tracked and summed.

The primary outcome will be the changes in total NSAID, opioid and acetaminophen use of the patients between the groups (rectus reapproximation and no rectus reapproximation groups). The investigators will also analyze the VAS scores of the patients 24 and 48 hours after surgery between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida pregnancies
* Singleton pregnancies
* Aged between 18- 45
* Term pregnancy
* First cesarean section
* Elective
* Without any comorbidity (Thyroid disorders, Diabetes Mellitus, Hypertension, Preterm delivery, etc.)

Exclusion Criteria:

* active labor,
* Prior cesarean section
* chronic analgesia use,
* vertical skin incision at cesarean,
* allergy to opioid or nonsteroidal anti-inflammatory drugs (NSAIDs),
* prior laparotomy,
* class III obesity (body mass index above 40).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Yes: Eligibility is based on gender
Study Population: This study is a prospective, randomized controlled trial conducted at Balikesir University, Department of Obstetrics and Gynecology at Balikesir Turkey. Pregnant women undergoing elective first cesarean section who were not in labor and consented to the trial were randomly assigned to receive rectus muscle reapproximation versus no reapproximation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | postoperative period first 48 hours.
  Drugs (mg)
Operation time | During operation
  Operation time: Hours
Changes in hemoglobin level | Intraoperative and postoperative period (including postoperative 48 hours)
  mg/dl
Length of hospital stay | Throughout postoperative period, an average of 2 days after surgery
  Length of hospital stay: Days
Occurence of postoperative complication | Throughout postoperative period, an average of 7 days after surgery
  Hematoma, dehiscense, blood transfusion, etc.
Postoperative pain | Visual analog score of the patient after 24 hours after cesarean section
  Visual Analog Scale Score: Units on a Scale (minimum score: 1- maximum score: 100)
Postoperative pain | Visual analog score of the patient after 48 hours after cesarean section
  Visual Analog Scale Score: Units on a Scale (minimum score: 1- maximum score: 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University Medical Faculty Department of Obstetrics and Gynecology, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.